CLINICAL TRIAL: NCT01045304
Title: Multicenter, Randomized, Open Label Study Evaluating a Poly(ADP-ribose) Polymerase-1(PARP-1) Inhibitor, SAR240550 (BSI-201), Administered Twice Weekly or Weekly, in Combination With Gemcitabine/Carboplatin, in Patients With Metastatic Triple Negative Breast Cancer (mTNBC)
Brief Title: Study of SAR240550 (BSI-201) in Combination With Gemcitabine/Carboplatin, in Patients With Metastatic Triple Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCD11418; 2009-016091-80 (EudraCT Number)
Record Dates: First submitted 2010-01-07; First posted 2010-01-11 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Breast Cancer, Metastatic
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — iniparib; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gencitabine + iniparib twice weekly (Experimental): Gemcitabine, 1000 mg/m² IV over 30 minutes and carboplatin, area under the curve (AUC) = 2, IV over 60 minutes, both on Days 1 and 8 of 3-week cycles.
  Iniparib, 5.6 mg/kg IV over 60 minutes on Days 1, 4, 8 and 11 of 3-week cycles
  Interventions: Drug: Iniparib; Drug: Gemcitabine; Drug: Carboplatin
- Gencitabine + iniparib weekly (Experimental): Gemcitabine, 1000 mg/m² IV over 30 minutes and carboplatin, area under the curve (AUC) = 2, IV over 60 minutes, both on Days 1 and 8 of 3-week cycles.
  Iniparib, 11.2 mg/kg IV over 60 minutes on Days 1 and 8 of 3-week cycles
  Interventions: Drug: Iniparib; Drug: Gemcitabine; Drug: Carboplatin

INTERVENTIONS:
Drug: Iniparib — Pharmaceutical form: solution for infusion
  Route of administration: intravenous
  Other Names: SAR240550; BSI-201
Drug: Gemcitabine — Pharmaceutical form: solution for infusion
  Route of administration: intravenous
Drug: Carboplatin — Pharmaceutical form: solution for infusion
  Route of administration: intravenous

SUMMARY:
Primary Objective:

* To assess the objective response rate (ORR) of iniparib (SAR240550) administered as a 60min intravenous (IV) infusion twice weekly or weekly, in combination with gemcitabine/carboplatin chemotherapy regimen in patients with metastatic Triple Negative Breast Cancer (mTNBC).

Secondary Objectives:

* To assess the clinical benefit rate (CBR) defined as the rate of complete response (CR), partial response (PR) and stable disease (SD) lasting at least 24 weeks;
* To assess Progression-free survival (PFS) and the overall survival (OS);
* To assess the safety profile of each schedule of iniparib;
* To assess the biological activity in tumor tissue (substudy);
* To evaluate the pharmacokinetic (PK) profile of iniparib (substudy);
* To characterize molecular and biological profile of tumors (substudy);
* To assess the effect of iniparib on poly(ADP)-ribose (PAR) level in peripheral blood mononuclear cells (PBMC) (substudy).

DETAILED DESCRIPTION:
The duration of the study for a patient includes a period for inclusion of up to 3 weeks. The patients may continue treatment until disease progression, unacceptable toxicity or consent withdrawal, followed by a minimum of 30-day follow-up after the last study treatment administration.

In case of discontinuation of study treatment, the patient will be considered as withdrawn from study treatment, and will be followed as planned for at least 30 days after the last administration of study treatment for safety purpose. In case of study treatment discontinuation without disease progression, efficacy data will be collected every 6 weeks until disease progression, death or end of study whatever comes first. After disease progression, the patient will be followed-up every 12 weeks (3 months) for overall survival until death or end of study.

The patients who benefit from the study treatment can continue until disease progression, toxicity or willingness to stop.

ELIGIBILITY:
Inclusion criteria:

* Histologically documented breast cancer (either primary or metastatic site) that is ER (estrogen receptor)-negative, PgR (progesterone receptor)-negative ( <10% tumor staining by immunohistochemistry [IHC]) and HER2 (human epidermal growth factor 2) non-overexpressing by IHC (0,1+) or, IHC 2+ and FISH (fluorescence In situ hybridization) negative.
* Metastatic breast cancer with measurable disease by the revised guideline for Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1 criteria);
* Prior treatment that includes:

  * never having received anticancer therapy for metastatic disease OR
  * having received 1 or 2 prior chemotherapy regimens in the metastatic setting (prior neo-adjuvant/adjuvant systemic therapy is considered as a prior chemotherapy if the first relapse occurred less than one year after the last treatment administration).

Exclusion criteria:

* Prior treatment with gemcitabine, carboplatin, cisplatin or any PARP inhibitor;
* Bone metastasis as only disease location (except for bone metastasis with measurable soft tissue component);
* Major medical conditions that might affect study participation e.g., uncontrolled pulmonary, renal, or hepatic dysfunction, uncontrolled infection, cardiac disease.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2010-02; Primary Completion 2011-03 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up the cut-off date for analysis defined as 16 weeks after the 1st dose in the last participant (maximum follow-up of 14 months)
  Proportion of participants with confirmed complete response (CR) or partial response (PR) as confirmed by an Independent Radiology Review Committee (IRRC) based on central review of scans in a blinded manner.

SECONDARY OUTCOMES:
Clinical benefit rate (CBR) | Up the cut-off date for analysis defined as 16 weeks after the 1st dose in the last participant (maximum follow-up of 14 months)
  Proportion of participants with confirmed complete response (CR) or partial response (PR) ot stable disease (SD) greater than 24 weeks as confirmed by the IRRC.
Progression-free survival | Up the cut-off date for analysis defined as 16 weeks after the 1st dose in the last participant (maximum follow-up of 14 months)
  Number of days from the date of randomization to the date of disease progression (ie, radiological progression based on IRRC assessment) or the date of death (from any cause), whichever is earlier.
Overall survival | Up the cut-off date for analysis defined as 16 weeks after the 1st dose in the last participant (maximum follow-up of 14 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (20):
- Australia (3):
  - Sanofi-Aventis Investigational Site Number 036002, Parkville
  - Sanofi-Aventis Investigational Site Number 036001, Perth
  - Sanofi-Aventis Investigational Site Number 036003, Westmead
- Belgium (2):
  - Sanofi-Aventis Investigational Site Number 056001, Brussels
  - Sanofi-Aventis Investigational Site Number 056002, Leuven
- France (6):
  - Sanofi-Aventis Investigational Site Number 250005, Besançon
  - Sanofi-Aventis Investigational Site Number 250003, Bordeaux
  - Sanofi-Aventis Investigational Site Number 250002, Dijon
  - Sanofi-Aventis Investigational Site Number 250006, Paris
  - Sanofi-Aventis Investigational Site Number 250004, Paris
  - Sanofi-Aventis Investigational Site Number 250001, Toulouse
- Italy (4):
  - Sanofi-Aventis Investigational Site Number 380004, Genova
  - Sanofi-Aventis Investigational Site Number 380001, Milan
  - Sanofi-Aventis Investigational Site Number 380002, Modena
  - Sanofi-Aventis Investigational Site Number 380003, Udine
- Sanofi-Aventis Investigational Site Number 528001, Rotterdam, Netherlands
- Spain (4):
  - Sanofi-Aventis Investigational Site Number 724002, Barcelona
  - Sanofi-Aventis Investigational Site Number 724004, Madrid
  - Sanofi-Aventis Investigational Site Number 724001, Málaga
  - Sanofi-Aventis Investigational Site Number 724003, Valencia

REFERENCES:
- [Derived] Dieras V, Bonnefoi H, Alba E, Awada A, Coudert B, Pivot X, Gligorov J, Jager A, Zambelli S, Lindeman GJ, Charpentier E, Emmons GT, Garcia-Ribas I, Paridaens R, Verweij J. Iniparib administered weekly or twice-weekly in combination with gemcitabine/carboplatin in patients with metastatic triple-negative breast cancer: a phase II randomized open-label study with pharmacokinetics. Breast Cancer Res Treat. 2019 Sep;177(2):383-393. doi: 10.1007/s10549-019-05305-w. Epub 2019 Jun 6. PMID 31172407